CLINICAL TRIAL: NCT00853528
Title: Cyberknife Radiosurgery for Improving Palliation of Metastatic Tumors of the Spine
Brief Title: Stereotactic Radiosurgery in Treating Patients With Spinal Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Minh Tam Truong, BMC Attending Physician, Boston Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26577; W81XWH-07-1-0342 (Other Grant/Funding Number: Dept of Defense); CDR0000635267 (Other: BUMC)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Cancer
Keywords: spinal cord metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Intervention Model Description: This is a Phase I study with 2 parallel groups of dose escalation using a 3 +3 design to determine the maximum tolerated dose of the radiation with the FDA approved device. There are three dose cohorts in each group, thus 6 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Single-fraction radiosurgery; 16 Gray (Experimental): Subjects able to achieve the spinal cord dose constraints for single-fraction SRS stereotactic radiosurgery Radiation: stereotactic radiotherapy at 16 Gray Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: single-fraction SRS
- Hypo-fractionated radiosurgery; 21 Gray (Experimental): Subjects unable to achieve the spinal cord dose constraints for single-fraction radiosurgery (SRS), based on tumor location and expected tolerance dose to the adjacent normal tissue, will be offered hypo-fractionated SRS (3 fractions) Radiation: stereotactic radiotherapy Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging hypo-fractionated radiation therapy at 21 Gray
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: hypo-fractionated SRS
- Single-fraction radiosurgery; 18 Gray (Experimental): Subjects able to achieve the spinal cord dose constraints for single-fraction SRS stereotactic radiosurgery Radiation: stereotactic radiotherapy at 18 Gray Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: single-fraction SRS
- Single-fraction radiosurgery; 20 Gray (Experimental): Subjects able to achieve the spinal cord dose constraints for single-fraction SRS stereotactic radiosurgery Radiation: stereotactic radiotherapy at 20 Gray Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: single-fraction SRS
- Hypo-fractionated radiosurgery; 24 Gray (Experimental): Subjects unable to achieve the spinal cord dose constraints for single-fraction radiosurgery (SRS), based on tumor location and expected tolerance dose to the adjacent normal tissue, will be offered hypo-fractionated SRS (3 fractions) Radiation: stereotactic radiotherapy Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging hypo-fractionated radiation therapy at 24 Gray
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: hypo-fractionated SRS
- Hypo-fractionated radiosurgery; 27 Gray (Experimental): Subjects unable to achieve the spinal cord dose constraints for single-fraction radiosurgery (SRS), based on tumor location and expected tolerance dose to the adjacent normal tissue, will be offered hypo-fractionated SRS (3 fractions) Radiation: stereotactic radiotherapy Questionnaire administration diffusion tensor imaging functional magnetic resonance imaging hypo-fractionated radiation therapy at 27 Gray
  Interventions: Other: questionnaire administration; Procedure: diffusion tensor imaging; Procedure: functional magnetic resonance imaging; Radiation: hypo-fractionated SRS

INTERVENTIONS:
Other: questionnaire administration — prior to radiosurgery, at radiosurgery completion, and then at subsequent follow-ups (3, 6, 9, 12, 18, and 24 months after treatment
Procedure: diffusion tensor imaging — prior to initiating CyberKnife radiosurgery, at 6 weeks after CyberKnife therapy, and at 6 months after CyberKnife therapy
Procedure: functional magnetic resonance imaging — prior to CyberKnife, at 6 weeks, and 3 months after CyberKnife?, every 3 months for the first year, and every 6 months thereafter
Radiation: hypo-fractionated SRS — two to three consecutive daily sessions within one week for 3 cohorts- Cohort 1 = 21 Gy; Cohort 2 = 24 Gy; Cohort 3 = 27 Gy
  Arms: Hypo-fractionated radiosurgery; 21 Gray; Hypo-fractionated radiosurgery; 24 Gray; Hypo-fractionated radiosurgery; 27 Gray
Radiation: single-fraction SRS — two to three consecutive daily sessions within one week for 3 cohorts- for 3 cohorts- Cohort 1 = 16 Gy; Cohort 2 = 18 Gy; Cohort 3 = 20 Gy
  Arms: Single-fraction radiosurgery; 16 Gray; Single-fraction radiosurgery; 18 Gray; Single-fraction radiosurgery; 20 Gray

SUMMARY:
RATIONALE: Stereotactic radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue. It may also help patients with spinal metastases live more comfortably.

PURPOSE: This phase I trial is studying the side effects and best dose of stereotactic radiosurgery in treating patients with spinal metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To implement CyberKnife® technology for improving palliation in patients with spinal metastases.
* To determine the maximum tolerated dose of CyberKnife® hypofractionated stereotactic radiosurgery in these patients.
* To evaluate functional and diffusion MRI parameters in the spinal cord and tumor after treatment with Cyberknife® radiosurgery.

OUTLINE: Patients undergo placement of gold fiducial markers at the time of open surgical resection or percutaneous needle biopsy. Patients then undergo CyberKnife® hypofractionated stereotactic radiosurgery over 30-90 minutes daily for 2-3 days.

Patients undergo functional MRI and diffusion tensor imaging at baseline and then at 6 weeks and 6 months after completion of treatment. Patients also complete a pain questionnaire at baseline and then at 3, 6, 9, 12, 18, and 24 months after completion of treatment.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic spinal tumor

  * Localized spinal metastasis, defined as one of the following:

    * Solitary spinal metastasis
    * Two contiguous spinal levels

      * No more than 2 adjacent spinal levels involved by a single tumor
    * Involvement of ≤ 3 separate sites (e.g., C5, T5, and T12)
  * Tumor size ≤ 5 cm

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 6 months
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be ambulatory

Exclusion Criteria:

* Not pregnant or nursing
* No spinal instability
* No rapid neurological decline
* No bony retropulsions causing neurological abnormalities
* No total paraplegia for > 48 hours
* No psychological issues that would preclude completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for spinal tumor that would result in potential overlap of radiotherapy fields
* No treatment that is expected to exceed spinal cord tolerance or other regional normal tissue tolerance
* No tumors that are exquisitely radiosensitive and controlled with conventional radiotherapy (e.g., lymphoma, leukemia, multiple myeloma, or germ cell tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose - single fraction | 6 weeks
  Maximum tolerated dose of CyberKnife® hypofractionated stereotactic radiosurgery
Maximum tolerated dose - hypofraction | 6 weeks
  Maximum tolerated dose of CyberKnife® hypofractionated stereotactic radiosurgery

SECONDARY OUTCOMES:
Assessment of pain | baseline and then at 3, 6, 9, 12, 18, and 24 months after completion of treatment
  Pain as measured by the Brief Pain Inventory and Roland scale
Spinal cord response | baseline and then at 6 weeks and 6 months after completion of treatment
  Spinal cord response as measured by functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Tam Truong, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.